CLINICAL TRIAL: NCT03920306
Title: A Prospective Evaluation of Non-Operative Treatments for Gastrocutaneous Fistulae in Children
Acronym: GCF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Montreal Children's Hospital of the MUHC (Other); St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Robert Baird, Clinical Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H17-02821
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Gastrocutaneous Fistula; Gastrostomy Complications
Keywords: gastrostomy
MeSH Terms: interventions — Silver Nitrate; octyl 2-cyanoacrylate

STUDY DESIGN:
Intervention Model Description: Single prospective arm; historical control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Drug administration for the experimental arm includes:
  1. AgNO3 applied to the fistula tract.
  2. A topical adhesive of either 2-Octylcyanoacrylate glue (Dermabond), or Fibrin glue, or Histoacryl glue (Tissue Seal), will be applied over the fistula's aperture.
  3. Oral anti-reflux therapy of either Pantoprazole 20-40mg PO OD, or Ranitidine 5-10mg/kg/day PO divided twice daily or 150mg PO BID, for either 4 weeks or until gastrocutaneous fistula tract closure, whichever comes first.
  Interventions: Drug: oral anti-acid treatment

INTERVENTIONS:
Drug: oral anti-acid treatment — This study investigates a bundle of three commonly used treatments
  Other Names: Silver Nitrate; Dermabond

SUMMARY:
Gastrostomy tube placement is a common surgery, and involves placing a tube from the child's skin to the inside of their stomach, allowing an alternative route for nutrition and medication to patients who cannot tolerate oral intake. A common complication of gastrostomy tubes is the development of a persistent connection between the stomach and skin after their removal. This is called a gastrocutaneous fistula (GCF). Non-surgical options have shown some success in eliminating the need for surgery to close these fistulae. Their true efficacy is unknown however; this study evaluates a non-surgical intervention bundle in the prevention and treatment of GCFs.

DETAILED DESCRIPTION:
Purpose:To compare the efficacy of a non-surgical intervention bundle for the prevention and treatment of persistent gastrocutaneous fistulae.

Hypothesis: The investigators hypothesize that the bundled delivery of 3 non-surgical interventions will reduce the development of GCFs and subsequently the need for surgical closure as compared to an established historical control group.

Justification: Persistent gastrocutaneous fistulae are common complications after gastrostomy tube removal (33%), with the current gold-standard treatment being operative intervention; exposing the child to the risks of anesthesia and surgery. Several non-surgical treatments exist, and have shown promise in small retrospective studies, however their true efficacy is yet to be elucidated through a prospective trial. Non-surgical treatment options include the use of proton-pump inhibitors, topical fibrin glue, silver nitrate application, and collagen plugging. As standard of care, patients may receive one, none or a combination of these non-surgical treatments based on clinician decision.

Objectives: The objective of this study is to prospectively evaluate the efficacy of a bundled delivery of non-surgical adjuncts immediately after gastrostomy tube removal and compare outcomes to the historical rate of GCF development.

Research Design: This study is a prospective observational "pre-post" study, which will compare our intervention arm (non-surgical intervention bundle) with a recently established historical control group (completed systematic review of all reported cases). Baseline data will be entered at the time of enrollment. Assessment of our primary outcome (rate of GCF one month after treatment) and secondary outcomes (including an estimate of treatment cost, complications, treatment satisfaction, and need for further interventions) will be made at standard 2 and 4 week follow-up visits.

Statistical Analysis: Standardized quantitative hypothesis testing will be performed for the primary outcome with the aid of a local biostatistician. Power analysis has been established based on a 50% reduction in GCF development, with a sample size of 100 subjects. Secondary outcomes will be tabulated and subjected to quantitative or qualitative assessment as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for gastrostomy tube removal

Exclusion Criteria:

* Recurrent gastrocutaneous fistula
* Non-consenting
* Unable to comply with follow up assessments
* Known allergic reaction to study products

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Gastrocutaneous Fistula (GCF) | 1 month
  Rate of gastrocutaneous fistula persistence based on clinical assessment

OTHER OUTCOMES:
Caregiver satisfaction Survey | 1 month
  A 9 question Likert-style (Strongly disagree- Strongly agree) questionnaire evaluating caregiver perceptions of the study

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] St-Louis E, Safa N, Guadagno E, Baird R. Gastrocutaneous fistulae in children - A systematic review and meta-analysis of epidemiology and treatment options. J Pediatr Surg. 2018 May;53(5):946-958. doi: 10.1016/j.jpedsurg.2018.02.022. Epub 2018 Feb 8. PMID 29506816